CLINICAL TRIAL: NCT01161108
Title: A Randomized Controlled Trial Pilot Project to Evaluate the Efficacy of Melatonin in Children With Insomnia, Intractable Epilepsy and Neurodevelopmental Disabilities
Brief Title: Trial of Melatonin to Improve Sleep in Children With Epilepsy and Neurodevelopmental Disabilities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Shelly Weiss, Staff neurologist, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1000010842
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy; Insomnia; Developmental Disability
Keywords: Pediatrics; Epilepsy; Insomnia; Melatonin
MeSH Terms: conditions — Epilepsy; Sleep Initiation and Maintenance Disorders; Developmental Disabilities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: Fast Release Melatonin (Active Comparator): Subjects will be randomized to one of the two treatment arms and to the order of study medication v.s. placebo.
  The subject will undergo the assigned treatment for 7 weeks (3 weeks of study drug, a one week wash-out and 3 weeks of placebo, or vice versa).
  Interventions: Drug: Fast Release Melatonin (FR MLT); Drug: Fast Release Placebo
- Group B: Timed Release Melatonin (Active Comparator): Subjects will be randomized to one of the two treatment arms and to the order of study medication v.s. placebo.
  The subject will undergo the assigned treatment for 7 weeks (3 weeks of study drug, a one week wash-out and 3 weeks of placebo, or vice versa).
  Interventions: Drug: Timed Release Melatonin (TR MLT); Drug: Timed Release Placebo

INTERVENTIONS:
Drug: Fast Release Melatonin (FR MLT) — 3mg capsules of melatonin will be used. The dose of FR MLT will be 3 mg for children less than or equal to 20 kg, and 6 mg for children greater than 20 kg. The study medication will be given one hour before bedtime, once daily.
  Other Names: Sleep Tight TM by Nature's Harmony® Melatonin
  Arms: Group A: Fast Release Melatonin
Drug: Fast Release Placebo — A matching FR MLT placebo will be compounded by the SickKids research pharmacy.
  The dose of Fast Release Placebo will be 3 mg for children less than or equal to 20 kg, and 6 mg for children greater than 20 kg. The study medication will be given one hour before bedtime, once daily.
  Arms: Group A: Fast Release Melatonin
Drug: Timed Release Melatonin (TR MLT) — 3 mg capsules will be used.
  The dose of TR MLT will be will be 3 mg for children less than or equal to 20 kg, and 6 mg for children greater than 20 kg. The study medication will be given one hour before bedtime, once daily.
  Other Names: Melatonin Timed Release by General Nutrition Canada
  Arms: Group B: Timed Release Melatonin
Drug: Timed Release Placebo — A matching TR MLT placebo will be compounded by the SickKids research pharmacy.
  The dose of Timed Release Placebo will be will be 3 mg for children less than or equal to 20 kg, and 6 mg for children greater than 20 kg. The study medication will be given one hour before bedtime, once daily.
  Arms: Group B: Timed Release Melatonin

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of oral melatonin in improving sleep continuity in children with epilepsy and neurodevelopmental delay who have chronic insomnia by comparing Fast Release Melatonin (FR MLT) to placebo and Timed Release Melatonin (TR MLT) with placebo in a randomized cross-over design trial.

DETAILED DESCRIPTION:
Sleep disturbance in children is a universal concern. The prevalence of sleep disorders may be as high as 80% in children with neurodevelopmental disabilities. The majority of the parental complaints are with difficulty getting children to settle to sleep at night and stay asleep (insomnia).

Two recent studies comparing children with epilepsy to matched controls or to sibling controls both concluded that children with epilepsy have more daytime sleepiness that may be due to underlying sleep disorders, and significantly greater sleep problems than their non-epileptic peers.

Endogenous melatonin is thought to synchronize the sleep-wake pattern with the light-dark cycle of the normal day. Exogenous melatonin has been found to be effective in reducing sleep onset latency, increasing sleep duration, and increasing sleep efficiency in a meta-analysis of subjects with sleep disorders. The melatonin in fast release preparations is released quickly and has a short half-life of less than 1 hour. It is most helpful in decreasing sleep onset latency (the time to fall asleep). The melatonin in timed release tablets is released in a slower more sustained way and, in a small study in children with severe neurodevelopmental disabilities, was more useful for sleep maintenance.

Fast release melatonin has been shown to be effective in a study of children with multiple disabilities and in one trial in children with epilepsy. Further rigorous evaluation of melatonin is needed as the validity of these studies is limited by their lack of blinding, small sample sizes, and subjective methods of sleep-wake outcome evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-17 years
* Children with epilepsy with at least 2 partial or generalized seizures per month over the last 3 months prior to starting the trial
* Children with neurodevelopmental disability, i.e. significant delay in development requiring special educational setting or educational assistant
* Anti-epileptic drugs (AED's) expected to remain unchanged for duration of trial (14 weeks)
* Not currently using melatonin or any other medication for sleep Subjects will be eligible if they have previous use of melatonin as long as there is a washout period of at least 1 week. Similarly, children taking natural health products for sleep will be included as long as there is a 30 day washout period prior to study enrollment.
* Chronic insomnia - reported by parent(s) to include one of the following: sleep onset latency of greater than one hour, duration of sleep less than 8.5 hours per night with either/or both these problems occurring at least 3 nights per week and that have occurred 3 months prior to trial, or night wakings of more than 2 per night for same time period

Exclusion Criteria:

* Planned epilepsy surgery or change in AED's during treatment trial
* Sleep disturbances that are treatable such as obstructive sleep apnea
* Allergy or severe adverse effects to melatonin
* Allergy or severe adverse effects to any of the ingredients of the study product or placebo (e.g. lactose)
* Lactose intolerance
* Pregnant
* Breastfeeding
* Known liver disease
* Ketogenic diet
* Other drugs being used for sedation
* Immunosuppressive drugs
* Known blood clotting abnormalities or who are on anticoagulant therapy (e.g. warfarin, blood thinners)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in duration of nocturnal sleep time | Baseline, Weeks 9 and 13
  We will measure the sleep time between 7 pm and 9 am.
  The measures will be analyzed to determine the change from baseline and change between active treatment and placebo.

SECONDARY OUTCOMES:
Sleep onset latency | Baseline, Weeks 9 and 13
  We will measure the interval of time between lights out and the onset of sleep.
  The measures will be analyzed to determine the change from baseline and change between active treatment and placebo.
Sleep efficiency | Baseline, Weeks 9 and 13
  We will measure the time sleeping/time in bed between lights out at night and lights on in the morning.
  The measures will be analyzed to determine the change from baseline and change between active treatment and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Shelly Weiss, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada